CLINICAL TRIAL: NCT01603394
Title: A Phase 4 Multicenter, Open-Label, Pilot Study Of Pregabalin And Prediction Of Treatment Response In Patients With Postherpetic Neuralgia
Brief Title: Pilot Study Of Pregabalin And Prediction Of Treatment Response In Patients With Postherpetic Neuralgia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9001464
Record Dates: First submitted 2012-04-16; First posted 2012-05-22 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (300-600 mg/day; 150 mg/day starting dose) (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Pregabalin Capsules (150 mg - 600mg), Dose titration (4 weeks) and fixed dose (2 weeks) for a 6 week treatment period.

SUMMARY:
The primary objective is to explore whether sensory symptom cluster analysis is useful for predicting treatment response in Postherpetic Neuralgia.

DETAILED DESCRIPTION:
The study was stopped on 26 April 2013 due to feasibility issues (low enrollment) not safety. The overall risk-benefit of Lyrica has not changed at all due to termination of this trial. Only 9 of the 150 patients were enrolled into the trial, so we are unable to get adequate results from this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have pain present for more than 3 months after the healing of the herpes zoster skin rash.
* At screening (V1) and baseline (V2), subjects must have a score of >=4 on the Numeric Rating Scale for Pain (1 week recall period).
* At baseline (V2), at least 4 pain diaries must be completed satisfactorily within the last 7 days and the average pain score must be >=4.

Exclusion Criteria:

* Subjects having other severe pain that may confound assessment or self evaluation of the pain due to PHN.
* Neurolytic or neurosurgical therapy for Postherpetic Neuralgia
* Skin conditions in the affected dermatome that could alter sensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (4):
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Jekintown, Pennsylvania
- Austria (2):
  - Pfizer Investigational Site, Senftenberg, A-3541
  - Pfizer Investigational Site, Vienna
- Pfizer Investigational Site, Schwerin, Germany
- South Africa (2):
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Paarl, Western Cape

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001464&StudyName=Pilot%20Study%20Of%20Pregabalin%20And%20Prediction%20Of%20Treatment%20Response%20In%20Patients%20With%20Postherpetic%20Neuralgia%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants were screened, of which nine participants at five study centers in the following four countries: Austria (2), Germany (1), South Africa (1) and USA (1) were enrolled and received at least one dose of pregabalin during the study.
Pre-assignment Details: This was a Phase 4, open-label, pilot study of pregabalin and prediction of treatment response in post herpetic neuralgia (PHN) participants. The duration of the treatment period was 6 weeks (4 weeks dose optimization +2 weeks fixed dose), with a 1-week taper/placebo washout administered at the end of study.
Groups:
- Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose): During the first week of treatment, participants received the starting dose of pregabalin of 150 mg/day Participants were then optimized to a dose of 300, 450 or 600 mg/day pregabalin based on efficacy and tolerability at each weekly visit: V3 (Week 1), V4 (Week 2), V5 (Week 3) and V6 (Week 4).
Period: Overall Study
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 9
Age, Customized [Number; unit: Age at least 18 years] | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Daily Pain Diary (Numerical Rating Scale, NRS) Mean Pain Score at the End of the Study (Week 6).
Description: The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
Time Frame: Baseline, Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

2. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) at All Visits.
Description: NPSI: participant rated questionnaire to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]). Includes 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each of the relevant dimensions and a total score of 0-100. Higher score indicates a greater intensity of pain.
Time Frame: All visits
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Phenotypes Within the 30% and 50% Responder Groups at Baseline and Week 6.
Description: To explore whether sensory symptom cluster analysis is useful for predicting treatment response in paticipants with PHN, identification of the phenotype was initially required of all participants using three different approaches (with or without the baseline PHQ-8, GAD-7 Pain Related Sleep Interference Score Scale, PCS): 1. PainDETECT at baseline, 2. PainPREDICT at baseline, 3. NPSI at baseline. Then for each of the above phenotypes the distribution of the pregabalin responders (using 30% and 50%) were to be compared.
Time Frame: Baseline, Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 6/Early Termination.
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 6/Early Termination
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportions of Participants With >/=30% and >/=50% Pain Reduction Based on Daily Pain Diary at Baseline and Week 6.
Description: The daily pain diary consists of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants describe their pain during the previous 24 hours by choosing the appropriate number between 0 and 10. Self-assessment is performed daily at bedtime on a telephone via interactive voice response system (IVRS). The endpoint mean pain score is defined as the mean of the last 7 daily diary pain ratings while taking study medication in the open-label phase. Daily pain IVRS diaries were completed daily at bedtime from Visit 1 (Screening) through Visit 7/Early Termination. Participants were asked to complete their first IVRS daily at bedtime on the morning after Visit 1.
Time Frame: Baseline, Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

6. Secondary Outcome: Proportion of Participants Within Each Phenotype Group as Determined by Sensory Symptom Clustering Using the PainPREDICT, PainDETECT and Neuropathic Pain Symptom Inventory at Baseline and Week 6.
Description: To explore whether sensory symptom cluster analysis is useful for predicting treatment response in paticipants with PHN, identification of the phenotype was initially required of all participants using three different approaches (with or without the baseline PHQ-8, GAD-7 Pain Related Sleep Interference Score Scale, PCS): 1. PainDETECT at baseline, 2. PainPREDICT at baseline, 3. NPSI at baseline.
Time Frame: Baseline, Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8) at Baseline and Week 6; Generalized Anxiety Disorder-7 (GAD-7) at Screening, Visit 2 (Week 0) and Week 6/Early Termination.
Description: The PHQ-8 is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as 0 (not at all) to 3 (nearly every day). The PHQ-8 is a validated subset of the PHQ-9, which comprises the first 8 items of the measure. The GAD-7 is a 7-item questionnaire that assesses anxiety. Participants respond as to how each item applies to them on a 4 point response scale. The higher the score, the more severe the anxiety.
Time Frame: Screening, Visit 2 (Week 0) and Week 6/Early Termination
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

8. Secondary Outcome: Brief Pain Inventory (BPI sf) at Visit 2 (Week 0) and Week 6.
Description: The Brief Pain Inventory-Short Form (BPI-sf) consists of 5 questions. Questions 1, 2, 3, and 4 measure pain on an 11-point scale from 0 (no pain) to 10 (worst pain possible).
Time Frame: Visit 2 (Week 0), Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

9. Secondary Outcome: Patient Catastrophizing Scale (PCS) at Visit 2 (Week 0) and Week 6.
Description: The PCS is a 13-item self report instrument and requires a Grade 6 reading level and has been translated into 12 languages. It instructs participants to reflect on past experience of pain and indicate their experience using a 5-point scale. The PCS was designed for research on catastrophizing and pain experience. Catastrophizing is associated with heightened pain and is "an exaggerated negative mental set brought to bear during actual or anticipated painful experience." It is a multidimensional construct compromising elements of rumination, magnification, and helplessness and its factor structure has been replicated. It has a total score and three subscale scores (score range of 0-52).
Time Frame: Visit 2 (Week 0), Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

10. Secondary Outcome: Pain NRS Score; 1 Week Recall Period.
Description: as for outcome 1
Time Frame: 1 Week
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

11. Secondary Outcome: Short Form 12v2 Health Survey (SF 12v2) at Visit 2 (Week 0), and Week 6/Early Termination.
Description: The Short-Form 12 Health Survey (SF-12v2) is a self-administered, validated questionnaire that measures each of the following 8 health aspects: Physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception over the past week. Higher scores indicate a better health-related quality of life.
Time Frame: Visit 2 (Week 0), and Week 6/Early Termination
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline to End of the Study (Week 6) in the Daily Sleep Interference Diary (NRS) Mean Pain Score.
Description: The pain-related sleep interference item rating scale is scored on an 11-point numeric rating scale (NRS-Sleep). It is self-administered by the participant in order to rate how pain has interfered with their sleep during the past 24 hours, ranging from 0 (pain does not interfere with sleep) to 10 (completely interferes (unable to sleep due to pain). Participants are to describe how their pain has interfered with their sleep during the past 24 hours by choosing the appropriate number on the numeric rating scale.
Time Frame: Baseline, Week 6
Population: Only 9 of the 200 participants were enrolled into the trial, so we are unable to get adequate results from this study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs: The time the participant had taken at least one dose of study treatment through last participant visit. SAEs: The time the participant provides informed consent through and including 28 calendar days after the last administration of study treatment.
Description: The same event may appear as both an adverse event (AE) and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose)
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (300-600 mg/Day; 150 mg/Day Starting Dose) (N=9)
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Edema peripheral (General disorders) | 2
Fatigue (General disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Outcome measure PCS was removed in protocol amendment1. Study stopped due to low enrolment and not safety. Efficacy analyses were not performed; safety results are described. Overall risk-benefit of pregabalin has not changed due to trial termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.